CLINICAL TRIAL: NCT04209556
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PARALLEL-GROUP, PLACEBO-CONTROLLED STUDY WITH AN OPEN LABEL EXTENSION TO EVALUATE THE SAFETY AND EFFICACY OF PF-06826647 IN PARTICIPANTS WITH MODERATE TO SEVERE ULCERATIVE COLITIS
Brief Title: A Study To Evaluate The Safety And Efficacy Of PF-06826647 In Participants With Moderate To Severe Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn following a strategic portfolio re-prioritization.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2501003; 2019-003999-39 (EudraCT Number)
Record Dates: First submitted 2019-12-01; First posted 2019-12-24 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ropsacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06826647 100 mg once a day (QD) (Experimental): PF-06826647 100 mg once a day (QD)
  Interventions: Drug: PF-06826647 100 mg QD
- PF-06826647 300 mg QD (Experimental): PF-06826647 300 mg QD
  Interventions: Drug: PF-06826647 300 mg QD
- PF-06826647 600 mg QD (Experimental): PF-06826647 600 mg QD
  Interventions: Drug: PF-06826647 600 mg QD
- Open Label Extension, PF-06826647 400 mg QD (Experimental): PF-06826647 400 mg QD
  Interventions: Drug: PF-6826647 400 mg QD

INTERVENTIONS:
Drug: PF-06826647 100 mg QD — Investigational Product
  Arms: PF-06826647 100 mg once a day (QD)
Drug: PF-06826647 300 mg QD — Investigational Product
  Arms: PF-06826647 300 mg QD
Drug: PF-06826647 600 mg QD — Investigational Product
  Arms: PF-06826647 600 mg QD
Drug: Placebo — Matched Placebo
  Arms: Placebo
Drug: PF-6826647 400 mg QD — Investigational Product
  Arms: Open Label Extension, PF-06826647 400 mg QD

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of PF-06826647 in moderate to severe ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe UC as defined by a total Mayo score of ≥6, with a rectal bleeding subscore of ≥1 and an endoscopic subscore of ≥2;
* Participants must have inadequate response to, loss of response to, or intolerance to at least one conventional therapy for UC: Oral, intravascular, or intramuscular corticosteroids; Immunosuppressants (azathioprine [AZA], 6-MP, or methotrexate [MTX]); Anti-tumor necrosis factor (TNF) inhibitors (eg, infliximab, adalimumab, or golimumab); Anti-integrin inhibitors (eg, vedolizumab); JAK inhibitor (eg, tofacitinib); Anti-IL-12/IL-23 inhibitors (eg, ustekinumab).

Exclusion Criteria:

* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, and diverticular disease associated with colitis, or Crohn's disease
* Participants displaying clinical signs of fulminant colitis or toxic megacolon;
* Participants with evidence of colonic dysplasia, adenomas or neoplasia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2023-10-26 (Estimated); Study Completion 2023-10-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving endoscopic response | At Week 8
  Endoscopic response is defined by Mayo endoscopic index < 2
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) based on severity and withdrawals due to adverse events (AEs) | At Week 60
Number of Participants With Clinical Laboratory Abnormalities | At Week 60
  Following parameters will be analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Percentage of participants with clinically significant changes in Electrocardiogram (ECG) | At Week 60
  Clinical significant changes in ECG
Number of Participants With Categorical changes from baseline in Vital Signs Data | At Week 60
  Number of participants with increase from baseline in sitting SBP and DBP of greater than or equal to 30 mmHg at Week 60.

SECONDARY OUTCOMES:
Percentage of participants achieving clinical remission | At Week 8 and 60
  Clinical remission is defined by total Mayo score of ≤ 2 with no individual subscore of > 1
Percentage of participants achieving endoscopic remission | At Week 8 and 60
  Endoscopic remission is defined as Mayo endoscopic index of 0
Percentage of participants achieving mucosal healing | At Week 8 and 60
  Mucosal healing is defined as both total Mayo score and histologic index of ≤ 1.
Percentage of participants achieving clinical response | At Week 8 and 60
  Clinical response is defined as a decrease from baseline of at least 3 points in total Mayo score with at least 30% change, accompanied by at least one point decrease or absolute score of 0 or 1 in rectal bleeding subscore.
Mean change from baseline in partial Mayo score over time | Up to 60 weeks
Change from baseline in total Mayo score | At Week 8 and 60
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) based on severity and withdrawals due to adverse events (AEs) | At Week 8
Number of Participants With Clinical Laboratory Abnormalities | At Week 8
  Following parameters will be analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Percentage of participants with clinically significant changes in Electrocardiogram (ECG) | At Week 8
  Clinically significant changes from baseline in ECG (heart rate, QT, QTc, PR and QRS intervals)
Number of Participants With Categorical Vital Signs Data | At Week 8
  Number of participants with increase from baseline in sitting SBP and DBP of greater than or equal to 30 mmHg at Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (24):
  - Hope Clinical Research, Canoga Park, California
  - ADVA Clinical Research, Inglewood, California
  - Centinela Valley Endoscopy Center, Inglewood, California
  - Inglewood Imaging Center, Inglewood, California
  - Surinder Saini, M.D., Inc., Newport Beach, California
  - Renaissance Imaging Center (CT/Xray), Northridge, California
  - Valley Endoscopy Center (Colonoscopy/Flexible sigmoidoscopy), Tarzana, California
  - Saludmax Medical Corp., Miami, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Gastroenterology Consultants P.C., Roswell, Georgia
  - Internal Medicine Associates (c/o TrialSpark, Inc.), Merrillville, Indiana
  - Gastroenterology Associates of New Jersey, LLC (c/o TrialSpark, Inc.), Clifton, New Jersey
  - Physicians Ambulatory Surgery Center, LLC, dba Physicians Endoscopy Center, Houston, Texas
  - Houston Digestive Diseases Consultants, P.A., Houston, Texas
  - Memorial Hermann SW Surgery Center, Houston, Texas
  - Gastroenterology Consultants of San Antonio, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - South Texas Radiology Imaging Center, San Antonio, Texas
  - Sugar Lakes Family Practice, PA, Sugar Land, Texas
  - Gastroenterolgy Associates of Northern Virginia, Fairfax, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Fair Oaks Imaging Center- Reston Radiology Consultants, Fairfax, Virginia
  - Associates in Gastroenterology (c/o TrialSpark, inc), Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501003